CLINICAL TRIAL: NCT04934735
Title: The Effectiveness of Case-management Rehabilitation Intervention in Facilitating Return to Work and Maintenance of Employment After Myocardial Infarction: Results of a Randomized Controlled Trial
Brief Title: Case-management Rehabilitation Intervention in Facilitating Return to Work After Myocardial Infarction
Acronym: CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, Shlomo Moshe, Head of Occupational Department, Assuta Hospital Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2006038
Record Dates: First submitted 2021-06-08; First posted 2021-06-22 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Case Manager; Myocardial Infarction; Sick Leave; Return to Work
Keywords: Rehabilitation, return to work, maintenance of employment
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled trial was conducted among patients who underwent an uncomplicated acute MI. Two weeks after hospitalization patients were referred to an examination by a cardiologist (to obtain a standardized clinical examination for all participants). Following this examination, the patients were assigned to an intervention group and a control group using simple randomization based on a computer-generated random sequence of numbers.
  The main outcomes are the rate of return to work in each phase of the study (meaning after 6,12,18, and 24 months)
Who Masked: Participant
Masking Description: The intervention group received a complex case-management rehabilitation program (described below) and the control group received the standard care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group: received a complex case-management rehabilitation program (Active Comparator): The intervention group was followed at 6, 12, 18, 24 months after entering the study. The follow-up was conducted by the case manager for patients in the intervention group, and by a research assistant for patients in the control group. Medical data were retrieved from the computerized medical records in the relevant hospitals.
  Interventions: Procedure: Rehabilitation program group
- The control: group received the standard care (No Intervention): The control group received regular care.

INTERVENTIONS:
Procedure: Rehabilitation program group — The case-management rehabilitation program was conducted by a clinical social worker within the occupational medicine clinic and included several components:
  1. Intake by a case manager
  2. Referral to an occupational physician was within one week of the intake.
  3. Charting an occupational rehabilitation program and timing the RTW date
  4. Coordinating between the patients and their family, treating physicians, the employer, community services, and meeting with the patient's family - all on a needful basis.
  5. Provision of a guidance booklet for employers on the RTW of cardiac patients.
  6. The psychosocial intervention was tailored to the patient's emotional state, occupational needs, and specific requests.
  7. Intensive follow-up sessions aimed to ensure that the rehabilitation program was carried out as planned.
  Other Names: complex case-management rehabilitation program
  Arms: The intervention group: received a complex case-management rehabilitation program

SUMMARY:
Abstract Purpose: To study the long-term effectiveness of case-management rehabilitation intervention among patients after myocardial infarction (MI) compared with the current standard of care.

Methods: Participants were 151 patients who underwent uncomplicated MI and of which nearly all enrolled in a cardiac rehabilitation program. Patients were randomized into an intervention or control group and provided two years of follow-up data. The intervention, conducted within an occupational medicine clinic, started during hospitalization or immediately thereafter and continued for 2 years. It included: early referral to an occupational physician, charting an occupational intervention program, coordinating between the patient and relevant parties, psychosocial intervention, intensive follow-up sessions during the first 1.5 months, and more spaced interventions during the follow-up period. Outcome variables were: return to work within 6 months of hospitalization and maintenance of employment at one and two years of follow-up.

DETAILED DESCRIPTION:
The program was conducted by a clinical social worker within the OM clinic and included several components:

1. Intake by a CM covering information regarding the rehabilitating program, assessing the patients' perception of their illness and the impact of the event on their life and family. Also included were: familiarization with the patient's occupational background, assessment of motivation, expectations, perceived efficacy and difficulties concerning RTW, and the identification of areas of intervention. Referral to further evaluation and treatment by a psychologist/psychiatrist was up to the CM's discretion.
2. Referral to an OP was within one week of the intake.
3. Charting an occupational rehabilitation program and timing the RTW date, not later than 35 days from hospital discharge. Before their RTW date, patients were invited for an additional meeting with the CM to facilitate their readiness to RTW and make any necessary arrangements.
4. Coordinating between the patients and their family, treating physicians, the employer, community services, and meeting with the patient's family - all on a needful basis.
5. Provision of a guidance booklet for employers on the RTW of cardiac patients. Patients could read it by themselves and/or hand it to their employer.
6. The psychosocial intervention was tailored to the patient's emotional state, occupational needs, and specific requests. When needed, short-term (up to 4 sessions) psychotherapeutic treatment was provided to help alleviate anxiety and other debilitating concerns, illness misconceptions, family issues, and occupational wavering.
7. Intensive follow-up sessions aimed to ensure that the rehabilitation program was carried out as planned, were conducted 2-, 4-, and 6-weeks after the beginning of the psychosocial intervention.

Intervention during follow-up

1. Patients who had RTW within three months after discharge from the hospital, received follow-up calls as follows: two weeks from the start of the CM intervention, every two months during the first six months, and once every six months thereafter (as outlined above). If needed, one or more of the above interventions were applied.
2. Patients who had not RTW within six months after discharge, due to psychosocial or employer-related issues received up to 12 intensive intervention sessions, in which the relevant parties were involved. Upon successful RTW, the six months follow-up calls were resumed.
3. Patients who had not RTW after six months for the above reasons, and were assessed as having rehabilitation potential, were referred to the National Social Security rehabilitation services and were followed up monthly for one year. The CM intervention was ended for patients without rehabilitation potential. For both groups, follow-up calls continued for six months.

The study received ethical approval from the institutional review board, serial number 2006038.

Statistical analysis Results are presented as mean + standard deviation (SD) for continuous variables and as frequencies for categorical variables. Data were analyzed using the SPSS statistical package (Version 26, SPSS Inc., Chicago, IL). Student's t-test was used to test for a difference between the means of two groups on a continuous dependent variable. Chi-square test of homogeneity was used to test for a difference between two proportions. For small groups, it was replaced by Fisher's exact test.

A multiple logistic regression model was used to investigate the relationship between employment status (employed/unemployed) at one year and two years of follow-up and CM program participation. Adjustments were made for factors that were found in previous studies to be associated with vocational re-integration and that could have confounded the findings of this study. A list of the possible confounders is presented in Table 4. Significance was determined by p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Sex/Gender: Both males and females
* Age limits: Minimum Age: 25 years old; Maximum age: 57 years old
* Clinical diagnosis: Patients after acute myocardial infarction
* Occupational status: Patients that have been working before the myocardial infarction
* HMO membership: Members in Maccabi Healthcare Service (HMO in Israel)
* Sampling Method: A consecutive participant sampling took place. Each patient who fulfilled the study terms was invited to participate in the study

Exclusion Criteria:

* Age over 57 years old or less than 25 years old
* Clinical diagnosis: Patients who had not sustained acute myocardial infarction
* Occupational status: Not working 6 months prior to the acute myocardial infarction
* HMO membership: Non-members of Maccabi Healthcare Service (HMO in Israel).
* Consent to participate: Patients who have not agreed to participate in the study

Max Age: 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2008-06-30 (Actual); Study Completion 2011-08-31 (Actual)

PRIMARY OUTCOMES:
Participants' return-to-work rates within 6 months from hospital discharge | Up to 6 months from hospital discharge
  This outcome measures the percentage of participants in either study or control groups, who have returned to work within 6 months of hospital discharge. This time window represents the optimal return to work period for most cardiac patients and assesses the effectiveness of the intervention in supporting the return to work process.
Percentage of participants that maintained their employment at 12, 18, and 24 months of follow-up | Up to 24 months from hospital discharge
  This outcome measures the percentage of participants in either study or control groups that have maintained their employment over time after having returned to work.
  Since some participants may not be capable of maintaining their employment status despite having returned to work, this outcome represents the effectiveness and quality of the return to work process and assesses the contribution of the case manager in supporting the participants' overall return to work.

SECONDARY OUTCOMES:
Occupational status of employed patients (full-time vs. part-time) | Up to 24 months from hospital discharge
  This outcome measures the degree of employment (full vs. part-time) of participants that have returned to work after their myocardial event.
  Some participants are able to return to full-time work, others need their work hours accommodated - this measure provides more information on the employment status amongst those that have managed to return to work and the effectiveness of the case manager in supporting the return to full-time work.
Occupational status of employed patients (Same vs. different job) | Up to 24 months from hospital discharge
  This outcome measures whether participants that return to work, will do so to their previous jobs/occupation or whether to a different job/occupation.
  Some participants are able to maintain the same job/occupation, others require accommodations and/or restrictions - this measure provides more information on the employment status amongst those that have managed to return to work and the effect the case manager will have in supporting the return to the same job/occupation.

CONTACTS AND LOCATIONS:
Overall Officials: Melamed Shmuel, Ass. Prof., Study Chair — Tal Aviv University
Locations (1):
- ‪Shlomo Moshe‬, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: No
Owing to data privacy regulations, the raw data for this study cannot be shared.

REFERENCES:
- [Derived] Zack O, Melamed S, Silber H, Cinamon T, Levy D, Moshe S. The Effectiveness of Case-management Rehabilitation Intervention in Facilitating Return to Work and Maintenance of Employment After Myocardial Infarction: Results of a Randomized Controlled Trial. Clin Rehabil. 2022 Jun;36(6):753-766. doi: 10.1177/02692155221076826. Epub 2022 Feb 22. PMID 35191331